CLINICAL TRIAL: NCT03018886
Title: Diagnosis of Adult Growth Hormone Deficiency With Growth Hormone Releasing Hormone Plus Arginine Stimulation Test
Brief Title: Diagnosing Adult Growth Hormone Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, tuula pekkarinen, consulting endocrinologist, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 203/2001 and 502/2002
Record Dates: First submitted 2017-01-06; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy control subjects (Other): 126 healthy controls underwent the GHRH plus arginine stimulations test
  Interventions: Other: GHRH plus arginine test
- patients with suspected GH deficiency (Experimental): 34 patients with pituitary disease and suspicion of GH deficiency underwent the GHRH plus arginine test
  Interventions: Other: GHRH plus arginine test

INTERVENTIONS:
Other: GHRH plus arginine test — One ug/kg GHRH [GHRH(1-29), GEREF Serono, Italy] was administered as an iv bolus at time 0 min, followed by arginine (L-arginine monohydrochloride, Braun, Melsungen, Germany) 0.5 g/kg (max 30g9 over 30 min. Blood samples were drawn at -15,0,15,30,45,60,75,90 min.

SUMMARY:
The purpose of this study was to validate the growth hormone releasing hormone (GHRH) plus arginine (GHRH+arg) stimulation test and it´s cut-off limits for diagnosis of adult growth hormone deficiency using the growth hormone (GH) Immulite 2000 Xpi assay calibrated against the IS 98/574 from the World Health Organization. A specific aim was to study the effect of gender and age on the peak GH response in the GHRH+arg test

DETAILED DESCRIPTION:
Adult growth hormone deficiency (AGHD) is a clinical entity including increased abdominal fat mass, decreased muscle mass, low bone density and adverse effects on quality of life and cardiovascular morbidity. These signs are nonspecific, and accurate diagnosis with laboratory tests in needed.

The GHRH+arg test is used to diagnose AGHD, but the cut-off values vary based on controls used. At moment consensus cut-off criteria are BMI specific, but gender and age may also affect the GH response in the GHRH+arg.

ELIGIBILITY:
Inclusion Criteria:

for health patients:

1. age 20-60 years,
2. no symptoms indicative of disease.

for patients:

1. age 16-90 years
2. previous pituitary disease
3. suspicion of growth hormone deficiency

Exclusion Criteria:

for healthy controls:

1. pregnancy,
2. a known or suspected disease,
3. any symptoms indicating disease
4. use of medication

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2001-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Peak serum GH (ug/l) by Immulite 2000 Xpi | one year

SECONDARY OUTCOMES:
Serum insulin like growth hormone 1 (IGF-1) concentration | one year
Basal serum GH (ug/l) by Immulite 2000 Xpi | one year

CONTACTS AND LOCATIONS:
Overall Officials: Esa Hamalainen, MD, PhD, Study Director — Chief, Department of Clinical Chemistry, Helsinki University Hospital, Helsinki, Finland
Locations (1):
- Tuula Pekkarinen, Helsinki, Finland